CLINICAL TRIAL: NCT02778386
Title: Phase I Trial to Assess the Safety and Pharmacokinetics of a Single Ascending Dose (SAD) of N-Methanocarbathymidine (N-MCT) in Normal Volunteers
Brief Title: Evaluating the Safety and Plasma Levels of N-Methanocarbathymidine (N-MCT) in Normal Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: N&N Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: N-MCT 329-15
Record Dates: First submitted 2016-04-27; First posted 2016-05-19 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Toxicity
MeSH Terms: interventions — (north)-methanocarbathymidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 6 subjects, male & female will receive one dose each of 200 mg of N-Methanocarbathymidine orally in capsules. Each subject will be evaluated for any clinical signs of any toxicity.
  Interventions: Drug: N-Methanocarbathymidine
- Cohort 2 (Experimental): 6 subjects, male & female will receive one dose each of 400 mg of N-Methanocarbathymidine orally in capsules. Each subject will be evaluated for any clinical signs of any toxicity.
  Interventions: Drug: N-Methanocarbathymidine
- Cohort 3 (Experimental): 8 subjects, males and females, 6 subjects will receive one dose each 800 mg of N-Methanocarbathymidine orally in capsules and 2 will receive a placebo capsule. Each subject will be evaluated for any clinical signs of any toxicity.
  Interventions: Drug: N-Methanocarbathymidine; Other: Placebo Capsule
- Cohort 4 (Experimental): 8 subjects, males and females, 6 subjects will receive one dose each 1200 mg of N-Methanocarbathymidine orally in capsules and 2 will receive a placebo capsule. Each subject will be evaluated for any clinical signs of any toxicity.
  Interventions: Drug: N-Methanocarbathymidine; Other: Placebo Capsule

INTERVENTIONS:
Drug: N-Methanocarbathymidine — Patients will receive 200 mg, 400 mg, 800 mg or 1200 mg of N-Methanocarbathymidine administered orally on day 1 after subject's full screen for each cohort. Each dose will be completely evaluated for safety and pharmacokinetics. The doses of each cohort will be given after complete evaluation of the preceding cohort for any sign of toxicity. In the absence of no observed toxicity, the next cohort will be started in the normal subjects.
  Other Names: N-MCT; NN-001
Other: Placebo Capsule — Two patients in Cohort 3 & 4 will receive placebo capsules which is mannitol filled into size 0 capsules.
  Other Names: Placebo
  Arms: Cohort 3; Cohort 4

SUMMARY:
This Phase I evaluation of N-MCT in normal volunteers requires sequentially increased doses. At each dose level, the safety and pharmacokinetic will be measured. This Phase I trial will have the dose range of N-MCT from 200mg - 1200mg per patient.

DETAILED DESCRIPTION:
This is a Phase 1 trial evaluating the safety and pharmacokinetics of N-MCT administered orally as a single ascending dose. Healthy male and female (non-pregnant, non-lactating) subjects ages 18-45, will be consented and allowed to participate in the study if upon screening they meet the inclusion / exclusion criteria.

Subjects will be enrolled into one of four cohort groups sequentially. Each of the six subjects in each group will receive doses sequentially within 48 hours between each dose increase (ie, the second subject in a group will not receive a dose until 48 hours after the first subject received a dose).

Cohort 1 (6 subjects, male & female) will receive 200 mg, Cohort 2 (6 subjects, male & female) will receive 400 mg, Cohort 3 (8 subjects, males and females, 2 placebo, 6 treated) will receive 800 mg and Cohort 4 (8 subjects, males and females, 2 placebo, 6 treated) will receive 1200 mg of N-MCT.

Each cohort will be completed and the safety data evaluated prior to initiating the next cohort. All subjects will have plasma and urine samples evaluated for N-MCT.

The PI of the protocol and the IDMC will review safety data (AEs), safety labs, vital signs, and findings through Day 7 for Cohort 1 before enrolling subjects in Cohort 2. Cohort 2 data through Day 7 will be reviewed accordingly by the PI and IDMC before enrolling subjects in Cohort 3. Cohort 3 data through Day 7 will be reviewed by the PI and the IDMC before enrolling subjects in Cohort 4.

However, prior to dose escalation to a new cohort as described above, GHUCCTS IRB will review and approve, in expedited review, the IDMC report upon which the decision to escalate the dose to a new cohort is based.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all Inclusion Criteria to be included in the study:

1. Healthy men and women 18 to 45 years of age, inclusive
2. Ability to understand the consent process and study procedures
3. Informed consent obtained and signed
4. Comprehension of the protocol, as determined by the clinic personnel using a series of questions after explaining the procedures.
5. Subjects agree to be available for all study visits.
6. General good health, no current medical illness or clinically significant abnormal physical examination findings as determined by study physician investigators
7. Negative past or current history of herpes virus infections, or no current use of antiviral medications for the treatment of herpes virus infections
8. Negative serum pregnancy test at screening and a negative serum pregnancy test on the day of admission to the inpatient phase for all female subjects of child bearing potential.
9. Negative urine toxicology screen for marijuana, cocaine, opiates, amphetamines, phencyclidine, benzodiazepines, and barbiturates for screening and on the day of admission to the inpatient phase.
10. Negative urine toxicology screen for nicotine (Cotinine) for screening and on the day of admission to the inpatient phase.
11. Negative breath alcohol screen and agreement not to consume alcohol for the duration of the study.
12. Body mass index (BMI) greater than or equal to 18.5 kg/m2 and less than or equal to 29.9 kg/m2 [weight (kg)]/ [height (m)2].
13. Agreement by subjects with reproductive potential to use highly effective contraception as described in protocol Section 4.1.1.
14. Willingness to avoid strenuous exercise for at least 72 hours prior to initial study drug administration and during the study to Day 7 visit.

Note: Strenuous physical exercise includes long distance running > 5 km/day, weight lifting, or any physical activity to which the subject is not accustomed.

Exclusion Criteria:

* Subjects meeting any of the Exclusion Criteria at Baseline will be excluded from study participation.

  1. Medical conditions that preclude participation in the study as determined by the study physician investigators.

     Note: Condition that may preclude participation includes:

     1.1. Vital signs that are outside the ranges in the table below, measured after at least 10 minutes rest:

     Blood Pressure (BP) 90-140/55-90 mmHg Pulse Rate (PR) 50 100 beats/min Tympanic Temperature (T) less than or equal to 37.6ºC Respiration Rate (RR) 12 to 20 breaths/minute

     1.2. Current diagnosis of pulmonary disease 1.3. Current diagnosis of asthma, which has required use of asthma medications within the past year 1.4. History of or current diagnosis of diabetes mellitus 1.5. Autoimmune disorder, such as systemic lupus erythematosus, Wegener's granulomatosis, rheumatoid arthritis 1.6. History of malignancy except low-grade skin cancer (i.e., basal cell carcinoma which has been surgically cured) 1.7. Chronic renal, hepatic, or pulmonary disease or gastrointestinal tract condition that could interfere with the absorption of the study drug (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, cholecystectomy, irritable bowel syndrome, inflammatory bowel disease) 1.8. History of cardiac abnormalities including Wolff-Parkinson-White syndrome, dysrhythmias, or coronary artery disease 1.9. History of prolonged QT interval
  2. Clinically significant abnormal electrocardiogram (ECG) at screening in the judgment of the investigator.
  3. Screening laboratory values outside the acceptable low and upper limits unless deemed NCS by the principal investigator or sub-investigator.
  4. Positive serology results for Hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) or human immunodeficiency virus (HIV) antibodies
  5. Febrile illness with temperature documented >38°C within 7 days of dosing
  6. Pregnancy or breastfeeding
  7. Known hypersensitivity or allergic reaction(s) to study drug components, including ingredients present in the formulation and/or to other nucleoside analogue antiviral drugs.
  8. Have consumed any prohibited products or undergone any prohibited procedure listed in Table 3 within the indicated time frame.
  9. Lack of ability to fully understand the informed consent. This will be determined by the recruiter/interviewer after explaining the consent and observing the subject reading the consent.
  10. Use of any form of tobacco, including cigarette smoking, pipe smoking, oral tobacco, for 30 days before screening and for the duration of the study.
  11. Any specific condition that, in the judgment of the Investigator, precludes participation because it could affect subject safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The Safety and Tolerability of N-MCT Evaluated By The Sequential Review of Reported Adverse Events (AEs) and Changes from Baseline in Findings on Physical Examination, Vital Sign Measurements, and Safety Laboratory Tests | Day 1- Day 7
  The type, incidence, severity and relatedness to study drug of adverse events (AEs), and of abnormal findings on physical examination, vital sign measurements, and of safety laboratory tests (hematology, biochemistry, urinalysis) throughout the study period.

SECONDARY OUTCOMES:
Plasma Concentrations of N-MCT Measured Before and at Multiple Time Points After Oral administration | Pre-Dose (0.000), 0.250, 0.500,0.750, 1.000, 1.500, 2.000, 2.500, 3.000, 4.000, 6.000, 8.000, 12.000, 24.000 and 48.000 hours
  Plasma levels of N-MCT will be measured before and at multiple time points after the oral administration.
  Plasma drug concentrations will be obtained at the following time points: pre-dose (0.000), 0.250, 0.500,0.750, 1.000, 1.500, 2.000, 2.500, 3.000, 4.000, 6.000, 8.000, 12.000, 24.000 and 48.000 hours.
Urine Concentrations of N-MCT Measured Before and at Multiple Time Points | 0 - 4, 4 - 8, 8 - 12, and 12 - 24 hours post dose
  Urine concentrations of N-MCT will be measured before and at multiple time points after the oral administration. Pooled urine samples for the measurement of N-MCT concentration will be collected over the following intervals: 0 - 4, 4 - 8, 8 - 12, and 12 - 24 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Aquilur Rahman, PhD, Study Director — N&N Pharmaceuticals Inc.
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided